CLINICAL TRIAL: NCT04361929
Title: Pediatric Difficult Airway Prediction Using Ultrasonography
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Nassar,MD, Associate professor, Cairo University
Other Study IDs: MS-259-2019
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Difficult Intubation; Difficult Mask Ventilation
Keywords: Difficult airway; pediatric; Airway ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — The following ultrasound measurements will be assessed: DS-HB, HMDR, TT, TT-S, TW, EW, ET, DS-E, and DS-V.

SUMMARY:
Recognition of difficult airway is purported to be the most important factor in successful management of difficult airway. The incidence of difficult airway in pediatrics is much less than in adults; however, airway related complications can lead to hypoxic brain damage or even death especially in younger age groups as neonates and infants.The aim of this work is to evaluate the feasibility and accuracy of ultrasound measurements (hyomental distances, tongue measurements, and anterior neck soft tissue thickness at the level of hyoid bone, thyrohyoid membrane, and thyroid cartilage) in predicting difficult laryngoscopy and difficult mask ventilation in pediatric patients undergoing elective surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Gender both males and females
* ASA Class I and II
* Age 1month to 10 years
* Children undergoing elective surgery under general anaesthesia

Exclusion Criteria:

* congenital upper airway malformation,
* head and neck swellings,
* scars,
* radiation to the neck,
* tracheotomy,
* Neurosurgical or cardiac procedures
* ENT surgeries

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 584 consecutive pediatric patients, aged one month-10 years scheduled for elective surgery under general anesthesia will be included in the study.
Sampling Method: Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2020-04-26 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
The sensitivity of DS-HB to predict difficult laryngoscopy | 30 minutes
  The ability of DS-HB ultrasound measurement to predict difficult airway in pediatrics

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy, Cairo, Egypt